CLINICAL TRIAL: NCT01577225
Title: A Prospective, Open, Randomised Controlled Trial to Compare OPSITE Post-Op Visible Wound Dressings With Standard Therapy in the Treatment of Surgical Incisions.
Brief Title: OPSITE Post-Op Visible Wound Dressings in Treatment of Surgical Incisions
Acronym: OPOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew Medical (Shanghai) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT10/02
Record Dates: First submitted 2012-04-12; First posted 2012-04-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2013-04

CONDITIONS: Patients Undergoing Clean Surgery
Keywords: Clean surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPSITE Post-Op Visible (Experimental): Subject is randomized to OPSITE Post-Op Visible group or Tape&Gauze group. Dressing should be used right after surgery and changed as needed.
  Interventions: Device: OPSITE POST-OP VISIBLE
- Tape&Gauze (Active Comparator): Subject is randomized to OPSITE Post-Op Visible group or Tape&Gauze group. Tape and Gauze should be used right after surgery and changed as per routin practice.
  Interventions: Device: Tape and Gauze

INTERVENTIONS:
Device: OPSITE POST-OP VISIBLE — Patient will be treated with OPSITE POST-OP VISIBLE dressing up to 14 days post surgery
  Arms: OPSITE Post-Op Visible
Device: Tape and Gauze — Patient will be treated with tape and gauze up to 14 days post surgery
  Arms: Tape&Gauze

SUMMARY:
OPSITE Post-Op Visible is a tri-layer dressing made up of a low adherent wound contact layer, lattice shaped absorbent pad and a top film that is waterproof and a bacterial barrier and is coated with a water-based adhesive. The comparator is a standard care treatment regime comprising tape and gauze.

This study requires 100 eligible patients which will be recruited from the patients routinely see by the study investigators at each study site. Eligible patients will undergo surgery that results in a surgical wound of 27cm or less that is expected to have low or moderate levels of exudate and will have received at least one randomised study treatment. The primary objective is to compare OPOV and tape/gauze in terms of wear time per patient.

DETAILED DESCRIPTION:
OPSITE Post-Op Visible (OPOV) is a post-operative dressing that has been developed to protect the wound from bacteria in the environment and absorb blood or other fluid exuding from the wound. The honeycomb nature of the dressing pad allows direct visibility of the wound through the dressing, minimising the need to expose the wound to the environment and the patient to the trauma of a dressing change just for the clinician to inspect the wound. OPOV is unique in combining these features and offers a real benefit over other standard post-operative dressing regimes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing "clean surgery" in an operating room
* Patients whose wounds will be closed surgically and not left to heal by secondary intention.
* Patients who are in-patients and are expected to be so for at least 5 days or are willing to return to the site for dressing changes.
* Patients who are at least 18 years of age.Patients who understand the trial and are willing to consent to the trial
* Patients who are willing to attend the post-discharge follow-up assessment.
* Patients whose wounds are up to 27cm in length (as measured from end to end in a straight line)
* Patients whose wounds are expected to have low to moderate exudate.

Exclusion Criteria:

* Pregnant or lactating females
* Patients undergoing chemotherapy, radiation therapy or taking any medication which is known to adversely affect wound healing
* Patients with a known medical condition or status known to delay or prevent normal wound healing such as diabetes, HIV, collagen vascular disorders and primary immune disorders
* Patients with a known sensitivity to any components of the investigational products or other similar dressings/products
* Patients with a history of poor compliance with medical treatment
* Patients who have participated in the study and who healed or were withdrawn.
* Patients who are unable to understand the aims and objectives of the trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Average wear time per patient | 0-14 days after surgery
  Average wear time per patient = Sum of evaluation dressing wear times for a patient/number of dressing applications

SECONDARY OUTCOMES:
Dressing wear time | 0-14 days after surgery
  Dressing wear time will be summarised by centre, type of surgical procedure, location of incision, incision length (≤ / > median) and level of exudate at the previous assessment for each treatment and overall.
Infection | 0-30 days after surgery
  Whether or not the wound was infected and if yes, whether it was superficial incisional, deep incisional or organ/space will be summarised at each dressing change, final assessment and 30 day post-surgery follow up by treatment and overall.
Clinical signs of infection | 0-30 days after surgery
  Clinical signs of infection will be summarised at each dressing change and final assessment will be summarised by centre, type of surgical procedure, incision length (≤ / > median), treatment and overall.
Dehiscence | 0-14 days after surgery
  Incidence of dehiscence during the treatment period, during the follow up period and during the study period and whether incidence of dehiscence was related to infection will be summarised by centre, type of surgical procedure, incision length (≤ / > median), treatment and overall.
Exudate management | 0-14 days after surgery
  The level of secretion/exudate will be summarised at each dressing change, final assessment and 30 day post-surgery follow up by centre, treatment and overall.
Condition of the surrounding skin (under the dressing) | 0-14 days after surgery
  Condition of the surrounding skin will be summarised at each dressing change and final assessment by centre, treatment and overall.
Patient comfort | 0-14 days after surgery
  Whether the dressing was comfortable during wear will be summarised by treatment and overall.
Dressing removal parameters | 0-14 days after surgery
  The reasons for dressing change will be summarised by treatment and overall.
Dressing conformability | 0-14 days after surgery
  Whether the dressing conformed to the area around the incision site upon dressing application and at dressing assessments will be summarised by treatment and overall.
Ease of application and removal | 0-14 days after surgery
  Ease of dressing application and ease of dressing will be summarised by treatment and overall.
Wound visibility through the dressing (OPOV dressings only) | 0-14 days after surgery
  Wound visibility through the dressing will be summarised at each dressing change assessment by treatment and overall. Additionally, this will be summarised by the level of exudate/secretion at the previous assessment.
Wound closure | 0-30 days after surgery
  Wound closure by 30 day post-surgery follow up treatment will be summarised by centre, type of surgical procedure, location of incision, incision length (≤ / > median), treatment and overall.
Length of hospital stay | 0-14 days after surgery
  Length of hospital stay will be summarised by baseline terms for centre, type of surgical procedure, location of incision and incision length (≤ / > median) for each treatment and overall.
Complications | 0-30 days after surgery
  Additional procedures as a result of complications (due to infection, dehiscence, haematoma, other) will be summarised by treatment and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Bingfang Zeng, Study Chair — Shanghai 6th People's Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Beijing Jishuitan Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No